CLINICAL TRIAL: NCT03573297
Title: A Double-blind, Placebo-controlled, Randomized Withdrawal, Multicenter Clinical Trial Evaluating the Efficacy, Safety and Tolerability of Cariprazine in a Dose-reduction Paradigm in the Prevention of Relapse in Bipolar I Disorder Patients Whose Current Episode is Manic or Depressive, With or Without Mixed Features
Brief Title: A Cariprazine Study in the Prevention of Relapse in Bipolar I Disorder Patients Whose Current Episode is Manic or Depressive, With or Without Mixed Features
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGH-MD-25; 2017-000803-25 (EudraCT Number)
Record Dates: First submitted 2018-06-05; First posted 2018-06-29 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Bipolar I Disorder; Mania; Depression
MeSH Terms: conditions — Mania; Depression | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Double-Blind Cariprazine 3.0 mg/day (Experimental): Participants randomized to receive cariprazine 3.0 mg once daily (QD) for up to 39 weeks.
  Interventions: Drug: Cariprazine
- Double-Blind Cariprazine 1.5 mg/day (Experimental): Participants randomized to receive cariprazine 1.5 mg QD for up to 39 weeks.
  Interventions: Drug: Cariprazine
- Double-Blind Placebo (Placebo Comparator): Participants randomized to receive placebo QD for up to 39 weeks.
  Interventions: Drug: Placebo
- Open Label Treatment (Experimental): Participants started on cariprazine 1.5 mg QD, with a target dose of 3.0 mg QD, for up to 16 weeks.
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine — Cariprazine capsules, oral administration, once daily
  Arms: Double-Blind Cariprazine 1.5 mg/day; Double-Blind Cariprazine 3.0 mg/day; Open Label Treatment
Drug: Placebo — Matching placebo capsules, oral administration, once daily
  Arms: Double-Blind Placebo

SUMMARY:
1) To evaluate the efficacy and safety of cariprazine at a target dose of 3.0 mg/day compared with placebo in prevention of relapse in patients with bipolar I disorder whose current episode (i.e. index episode) is manic or depressive, with or without mixed features; 2) To evaluate the efficacy and safety of cariprazine at a target dose of 1.5 mg/day compared with placebo in prevention of relapse in patients with bipolar I disorder whose current episode (i.e. index episode) is manic or depressive, with or without mixed features who were initially stabilized on a target dose of 3.0 mg/day

ELIGIBILITY:
Inclusion Criteria:

* Currently meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for bipolar I disorder, and at least one of the following two criteria:
* Current episode manic, with or without mixed features, having a total Young Mania Rating Scale (YMRS) total score ≥ 20 and a score of at least 4 on 2 YMRS items (irritability, speech, content, or disruptive/aggressive behavior);
* OR current episode depressive, with or without mixed features, having a Montgomery-Asberg Depression Rating Scale (MADRS) total score ≥ 23 and a score of at least 3 on 2 MADRS items (apparent sadness, reported sadness, inner tension or inability to feel).

Exclusion Criteria:

* Four or more episodes of a mood disturbance within the 12 months before Visit 1;
* Diagnosis of another psychiatric disorder other than bipolar disorder with the exception of specific phobias.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (108):
- United States (46):
  - Woodland International Research Group /ID# 232932, Little Rock, Arkansas
  - Woodland Research Northwest, LLC /ID# 232982, Rogers, Arkansas
  - California Pharmaceutical Research Institute Inc. /ID# 232745, Anaheim, California
  - Advanced Research Center /ID# 233120, Anaheim, California
  - CI Trials /ID# 232642, Bellflower, California
  - Synexus Clinical Research US Inc. /ID# 232743, Cerritos, California
  - ATP Clinical Research, Inc /ID# 232979, Costa Mesa, California
  - ProScience Research Group /ID# 232945, Culver City, California
  - Collaborative Neuroscience Research - Orange County /ID# 233077, Garden Grove, California
  - Behavioral Research Specialists, LLC /ID# 232980, Glendale, California
  - Omega Clinical Trials LLC /ID# 233150, La Habra, California
  - Synergy San Diego /ID# 232740, Lemon Grove, California
  - Alliance for Research - Long Beach /ID# 232926, Long Beach, California
  - NRC Research Institute /ID# 232741, Orange, California
  - CNRI-San Diego /ID# 232748, San Diego, California
  - Artemis Institute for Clinical Research /ID# 233151, San Marcos, California
  - Artemis Institute for Clinical Research /ID# 233152, San Marcos, California
  - Collaborative Neuroscience Research LLC /ID# 232750, Torrance, California
  - Duplicate_MCB Clinical Research Centers LLC /ID# 232838, Colorado Springs, Colorado
  - Velocity Clinical Research - Hallandale Beach /ID# 232647, Hallandale, Florida
  - Research Centers of America - Hollywood FL /ID# 232649, Hollywood, Florida
  - CNS Healthcare - Jacksonville /ID# 233160, Jacksonville, Florida
  - Meridien Research /ID# 232941, Maitland, Florida
  - Miami Lakes Medical Research /ID# 232826, Miami Lakes, Florida
  - University of South Florida /ID# 233093, Tampa, Florida
  - Synexus Clinical Research, Inc /ID# 232950, Atlanta, Georgia
  - Atlanta Center for Medical Research /ID# 232832, Atlanta, Georgia
  - CenExcel iResearch LLC /ID# 233045, Decatur, Georgia
  - Atlanta Behavioral Research, LLC /ID# 232935, Dunwoody, Georgia
  - NeuroPsychiatric Research Practice & Associate LTD /ID# 232840, Winfield, Illinois
  - Louisiana Clinical Research /ID# 232685, Shreveport, Louisiana
  - CBH Health LLC /ID# 232699, Gaithersburg, Maryland
  - St. Charles Psychiatric Associates - Midwest Research Group /ID# 232709, Saint Charles, Missouri
  - Duplicate_Altea Research Institute /ID# 232784, Las Vegas, Nevada
  - Hassman Research Institute /ID# 233088, Berlin, New Jersey
  - Neurobehavioral Research Inc /ID# 232791, Cedarhurst, New York
  - New Hope Clinical Research Inc. /ID# 232716, Charlotte, North Carolina
  - Richard Weisler MD, PA & Assoc /ID# 233049, Raleigh, North Carolina
  - Clinical Inquest Center Ltd /ID# 233043, Beavercreek, Ohio
  - DUPLICATE_The Ohios State University Department of Psychiatry /ID# 232739, Columbus, Ohio
  - Midwest Clinical Research Center /ID# 232737, Dayton, Ohio
  - Sooner Clinical Research /ID# 232931, Oklahoma City, Oklahoma
  - Community Clinical Research Inc. /ID# 232672, Austin, Texas
  - Pillar Clinical Research LLC /ID# 232667, Richardson, Texas
  - Pillar Clinical Research LLC /ID# 232673, Richardson, Texas
  - Family Psychiatry of The Woodlands /ID# 232943, The Woodlands, Texas
- Bulgaria (9):
  - Mental Health Centre - Prof.Dr.Ivan Temkov-Burgas /ID# 232777, Burgas
  - State Psychiatry Hospital-Kardzhali; Third Male Department /ID# 232779, Kardzhali
  - MHAT Dr. Hristo Stambolski EOOD; Hospital Pharmacy /ID# 232893, Kazanlak
  - State Psychiatric Hospital - Lovech /ID# 232771, Lovech
  - Second Psychiatric Clinic for General Psychiatry and Addictions of UMHAT Dr. Geo /ID# 232773, Pleven
  - UMHAT Dr Georgi Stranski EAD /ID# 233105, Pleven
  - UMHAT Kanev /ID# 233101, Rousse
  - Clinic of Child Psychiatry St Nicolas /ID# 232925, Sofia
  - MHAT Targovishte /ID# 232942, Targovishte
- Malaysia (2):
  - Hospital Raja Permaisuri Bainun /ID# 233114, Ipoh, Perak
  - University Malaya Med Ctr /ID# 233108, Kuala Lumpur
- Poland (4):
  - Specjalistyczny Gabinet Lekarski /ID# 232702, Lublin, Lublin Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 232848, Gdansk, Pomeranian Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska Filip Rybakowski /ID# 233170, Poznan, Silesian Voivodeship
  - Poradnia Zdrowia Psychicznego /ID# 232878, Chełmno
- INSPIRA Clinical Research /ID# 232704, San Juan, Puerto Rico
- Russia (14):
  - Kazan State Medical University /ID# 233110, Kazan', Tatarstan, Respublika
  - Mental Health Research Centre /ID# 232864, Moscow
  - Clinical Psychiatry Hospital #1 of Nizhniy Novgorod /ID# 232946, Nizhny Novgorod
  - Orenburg Regional Clinical Psychiatric Hospital #1 /ID# 232933, Orenburg
  - State Public Institution of Healthcare Leningrad Regional Psychoneurology Dispen /ID# 232872, Roschino
  - St. Nicolas Psychiatric Hospital /ID# 232858, Saint Petersburg
  - St. Nicolas Psychiatric Hospital /ID# 232859, Saint Petersburg
  - National Medical Research Center of Psychiatry and Neurology n.a. V.M. Bekhterev /ID# 232927, Saint Petersburg
  - National Medical Research Center of Psychiatry and Neurology n.a. V.M. Bekhterev /ID# 232928, Saint Petersburg
  - I. I. Skvortsov-Stepanov Psychiatric Hospital #3 /ID# 232930, Saint Petersburg
  - Saratov City Clinical Hospital #2 n.a. V. I. Razumovsky /ID# 232936, Saratov
  - Regional Clinical Psychiatry Hospital /ID# 232856, Saratov
  - Ltd Clinic Hundred Years /ID# 232866, Tomsk
  - Region Specialized Psychiatric Hospital #2 /ID# 232850, Tonnelniy
- Serbia (8):
  - University Clinical Center Serbia /ID# 233095, Belgrade, Beograd
  - University Clinical Center Kragujevac /ID# 233096, Kragujevac, Sumadijski Okrug
  - Clinical Center Vojvodina /ID# 233038, Novi Sad, Vojvodina
  - Clinical Hospital Center Dr Dragisa Misovic - Dedinje /ID# 232641, Belgrade
  - Institute of Mental Health /ID# 232958, Belgrade
  - Special Hospital for Psychiatric Diseases Kovin /ID# 232829, Kovin
  - Clinical Centre Kragujevac /ID# 232874, Kragujevac
  - Specialized Hospital for Neuropsychiatric Diseases Sveti Vracevi /ID# 232846, Novi Kneževac
- South Korea (5):
  - Inje University Busan Paik Hospital /ID# 233097, Busan
  - Inje University Haeundae Hospital /ID# 233141, Busan
  - Chonnam National University Hospital /ID# 233098, Gwangju
  - Jeju National University Hospital /ID# 233104, Jeju City
  - Duplicate_Chonbuk National University Hospital /ID# 232654, Jeonju
- Taiwan (5):
  - Taipei Veterans General Hospital /ID# 232947, Taipei City, Taipei
  - Taipei Tzu Chi Hospital /ID# 233128, New Taipei City
  - China Medical University Hospital /ID# 233091, Taichung
  - National Cheng Kung University Hospital /ID# 233109, Tainan
  - Tri-Service General Hospital /ID# 233078, Taipei
- Thailand (2):
  - Maharaj Nakorn Chiang Mai Hospital /ID# 232860, Chiang Mai
  - Suan Prung Psychiatric Hospital /ID# 232862, Muang
- Ukraine (12):
  - Cherkasy regional psychiatric hospital of the CRC /ID# 232686, Smila, Cherkasy Oblast
  - Geikivka multidisciplinary hospital for psychiatric care /ID# 232678, Kryvbas Village, Dnipropetrovsk Oblast
  - SI Institution Neurology Psychiatry and Narcology NAMS of Ukraine /ID# 232937, Kharkiv, Kharkivs’ka Oblast’
  - SI Institution Neurology Psychiatry and Narcology NAMS of Ukraine /ID# 232938, Kharkiv, Kharkivs’ka Oblast’
  - SI Institution Neurology Psychiatry and Narcology NAMS of Ukraine /ID# 232939, Kharkiv, Kharkivs’ka Oblast’
  - Kherson Regional Psychiatric Institution for Psychiatric Care /ID# 232684, Stepanivka Village, Kherson Oblast
  - Odesa regional psychiatric hospital 2 of the ORC /ID# 232682, Oleksandrivka Village, Odesa Oblast
  - KNP Zakarpatskyi Regional MC of Mental Health and Medicine of Dependencies /ID# 232680, Uzhhorod, Zakarpattia Oblast
  - Communal Institution of Lviv Regional Council Lviv Regional Clinical Psychiatric /ID# 232876, Lviv
  - MNCE Odesa Regional Medical Center for Mental Health /ID# 232944, Odesa
  - CI O.I. Yuschenko VRPsH Depts No.14 and No.15 M.I. Pyrogov VNMU /ID# 232853, Vinnytsia
  - Vinnytsia Regional Psycho-Neurological Hospital /ID# 232852, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 901 participants were enrolled; 5 participants did not enter the open label treatment period.
Groups:
- Open Label Treatment Period: Participants started on cariprazine 1.5 mg once daily (QD), with a target dose of 3.0 mg QD, for up to 16 weeks.
- Double-Blind Placebo QD: Partcipants randomized to receive placebo QD for up to 39 weeks.
- Double-Blind Cariprazine 1.5 mg QD: Participants randomized to receive cariprazine 1.5 mg QD for up to 39 weeks.
- Double-Blind Cariprazine 3.0 mg QD: Participants randomized to receive cariprazine 3.0 mg QD for up to 39 weeks.
Period: Open Label Treatment Period
Arm/Group | Open Label Treatment Period | Double-Blind Placebo QD | Double-Blind Cariprazine 1.5 mg QD | Double-Blind Cariprazine 3.0 mg QD
Started (Treated) | 896 | 0 | 0 | 0
Completed | 440 | 0 | 0 | 0
Not Completed | 456 | 0 | 0 | 0
Not completed — Adverse Event | 67 | 0 | 0 | 0
Not completed — Lack of Efficacy | 35 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 104 | 0 | 0 | 0
Not completed — Lost to Follow-up | 55 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 17 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 25 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 2 | 0 | 0 | 0
Not completed — Failure to Meet Randomization Criteria | 143 | 0 | 0 | 0
Not completed — Other, Not Specified | 7 | 0 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | Open Label Treatment Period | Double-Blind Placebo QD | Double-Blind Cariprazine 1.5 mg QD | Double-Blind Cariprazine 3.0 mg QD
Started (Randomized into Double-Blind Period) | 0 | 145 | 147 | 148
Randomized and Treated in Double-Blind Treatment Period | 0 | 145 | 144 | 147
Completed | 0 | 79 | 82 | 84
Not Completed | 0 | 66 | 65 | 64
Not completed — Relapse Event during Double-blind Treatment Period | 0 | 29 | 25 | 26
Not completed — Adverse Event | 0 | 1 | 5 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 23 | 11 | 14
Not completed — Lost to Follow-up | 0 | 4 | 4 | 9
Not completed — Protocol Violation | 0 | 3 | 8 | 4
Not completed — Non-Compliance With Study Drug | 0 | 0 | 4 | 4
Not completed — Other, Not Specified | 0 | 5 | 8 | 6

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least 1 dose of study medication.
Groups:
- Open Label Treatment Period: Participants started on cariprazine 1.5 mg QD, with a target dose of 3.0 mg QD, for up to 16 weeks.
Arm/Group | Open Label Treatment Period
Number analyzed (Participants) | 896
Age, Customized [Count of Participants; unit: Participants]
  < 45 years | 539
  ≥ 45 years | 357
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 542
  Male | 354
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 89
  Not Hispanic or Latino | 806
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 32
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 258
  White | 591
  More than one race | 10
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse of Any Mood Episode During the Double-Blind Treatment Period
Description: Relapse was defined as the occurrence of any 1 of the following:
  * Young Mania Rating Score (YMRS) total score ≥ 17 (range 0-60; higher score indicates a worse outcome);
  * Montgomery Asberg Depression Rating Scale; (MADRS) total score ≥ 20 (range 0-60; higher score indicates more depressive symptoms);
  * Clinical Global Impression-Improvement scale (CGI-S) ≥ 4 (range from 1 [normal, not at all ill] to 7 [extremely ill]);
  * Initiation of additional psychiatric medication;
  * Psychiatric hospitalization;
  * Exacerbation of illness as judged by clinical impression of the Investigator.
  Time to first relapse (days) was calculated as the date of the first relapse - the date of randomization + 1. Participants who did not meet the relapse criteria were considered censored at the time of completion or discontinuation from the Double-Blind Treatment Period (DBTP) of the study. Percentiles (95% Confidence Intervals [CI]) are based on Kaplan-Meier estimates.
Time Frame: From Week 16 to Week 55
Population: Double-Blind Intent-to-Treat Population: All participants who took at least 1 dose of DB IP and had at least 1 post-randomization assessment of the YMRS, MADRS or CGI-S scores or relapsed during the 39-week DBTP of the study.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Double-Blind Placebo QD: Participants randomized to receive placebo QD for up to 39 weeks.
Arm/Group | Double-Blind Placebo QD | Double-Blind Cariprazine 1.5 mg QD | Double-Blind Cariprazine 3.0 mg QD
Number analyzed (Participants) | 142 | 143 | 145
days
  25% percentile | NA [156.0 to NA] — Not estimable because the 3 treatment curves did not pass through the 25% percentile mark. | NA [220.0 to NA] — Not estimable because the 3 treatment curves did not pass through the 25% percentile mark. | NA [224.0 to NA] — Not estimable because the 3 treatment curves did not pass through the 25% percentile mark.
  50% percentile | NA [NA to NA] — Not estimable because the 3 treatment curves did not pass through the 50% percentile mark. | NA [NA to NA] — Not estimable because the 3 treatment curves did not pass through the 50% percentile mark. | NA [NA to NA] — Not estimable because the 3 treatment curves did not pass through the 50% percentile mark.
  75% percentile | NA [NA to NA] — Not estimable because the 3 treatment curves did not pass through the 75% percentile mark. | NA [NA to NA] — Not estimable because the 3 treatment curves did not pass through the 75% percentile mark. | NA [NA to NA] — Not estimable because the 3 treatment curves did not pass through the 75% percentile mark.
Statistical Analysis 1: Comparison: Double-Blind Placebo QD vs Double-Blind Cariprazine 1.5 mg QD; Test type: Superiority; p = 0.5745, Log Rank — P-value is based on the log-rank test stratified by modified index episode (manic or depressive) and region (US, non-US); Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.48 to 1.43] — Hazard ratio (Cariprazine 1.5 or 3.0 mg/day vs. Placebo) is based on Cox proportional hazards regression model, with treatment group as an explanatory variable, stratified by modified index episode (manic or depressive) and region (US, non-US)
Statistical Analysis 2: Comparison: Double-Blind Placebo QD vs Double-Blind Cariprazine 3.0 mg QD; Test type: Superiority; p = 0.6308, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.52 to 1.51] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Open Label Treatment Period: from enrollment (all-cause mortality [ACM]) or first dose of study drug (adverse events [AEs]) through Week 16 (Day113). Double-Blind Treatment Period (ACM/AEs): From first dose of double-blind treatment up to end of study, Week 59 (Day 414).
Description: ACM data include all enrolled (Open Label Treatment Period) or randomized (Double Blind Treatment Period) participants; AE data include all participants who were treated (Open Label Treatment Period) or randomized and treated (Double Blind Treatment Period).
Arm/Group | Open Label Treatment Period | Double-Blind Placebo QD | Double-Blind Cariprazine 1.5 mg QD | Double-Blind Cariprazine 3.0 mg QD
All-Cause Mortality (participants affected / at risk) | 1/901 | 1/145 | 0/147 | 0/148
Serious Adverse Events (participants affected / at risk) | 19/896 | 5/145 | 7/144 | 3/147
Other Adverse Events (participants affected / at risk) | 256/896 | 27/145 | 34/144 | 34/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment Period (N=896) | Double-Blind Placebo QD (N=145) | Double-Blind Cariprazine 1.5 mg QD (N=144) | Double-Blind Cariprazine 3.0 mg QD (N=147)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CORONAVIRUS PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SACRAL RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
BIPOLAR I DISORDER (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MANIA (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment Period (N=896) | Double-Blind Placebo QD (N=145) | Double-Blind Cariprazine 1.5 mg QD (N=144) | Double-Blind Cariprazine 3.0 mg QD (N=147)
NAUSEA (Gastrointestinal disorders) | 62 (64) | 1 (1) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8) | 4 (6) | 3 (3) | 10 (10)
WEIGHT INCREASED (Investigations) | 40 (40) | 7 (7) | 11 (12) | 13 (17)
AKATHISIA (Nervous system disorders) | 105 (117) | 2 (2) | 6 (7) | 2 (2)
HEADACHE (Nervous system disorders) | 79 (90) | 15 (22) | 14 (23) | 10 (13)
INSOMNIA (Psychiatric disorders) | 77 (85) | 5 (7) | 9 (12) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT03573297/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT03573297/SAP_001.pdf